CLINICAL TRIAL: NCT05449340
Title: Multidisciplinary Care Pathway With Electronic Patient Reported Outcomes (ePRO) Post-operative Follow-up of Breast Cancer Surgery Complications to Optimize Patient Quality of Life
Acronym: BEAUTIFY-3
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Prix Ruban Rose/2020/FF-03
Record Dates: First submitted 2022-06-27; First posted 2022-07-08 (Actual); Last update posted 2024-03-01 (Actual); Status verified 2024-02

CONDITIONS: Breast Cancer
Keywords: mastectomy; quality of life
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BEAUTIFY application (Experimental)
  Interventions: Device: BEAUTIFY application

INTERVENTIONS:
Device: BEAUTIFY application — Interview with the coordinating nurse in the postoperative period to install the BEAUTIFY application on the patient's smartphone and to train her to record any Patients will monitor their symptoms weekly. In case of toxicity grade > 2, the nurse will contact the patient for further information.

SUMMARY:
This project is a follow-on study of the BEAUTIFY-2 study (NCT04957186). The "BEAUTIFY" (BrEast cAncer qUaliTy of lIfe aFter surgerY) program was built by a committee of experts on the basis of reflections carried out within 2 focus groups. An application was developed to track patient reported outcome measures.

The study investigators now wish to evaluate the feasibility and impact on pain and quality of life of the "BEAUTIFY" care pathway on a larger cohort. The study hypothesis is that multidisciplinary care organization will improve the management and the quality of life post-breast cancer surgery.

ELIGIBILITY:
Inclusion Criteria:

* Breast cancer patient scheduled for surgery
* Patient able to use a connected electronic object and having a tablet or a smartphone with internet access at home.
* The patient must have given their free and informed consent and signed the consent form
* The patient must be a member or beneficiary of a health insurance plan

Exclusion Criteria:

* The subject is participating in a category 1 interventional study, or is in a period of exclusion determined by a previous study
* The subject unable to express consent
* It is impossible to give the subject informed information
* The patient is under safeguard of justice or state guardianship

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2022-07-25 (Actual); Primary Completion 2024-02-16 (Actual); Study Completion 2024-02-16 (Actual)

PRIMARY OUTCOMES:
Patient compliance with the program | End of study (12 months)
  Yes/No: study will be considered feasible if at least 80% of patients complete the program
Patient satisfaction with the intervention | End of study (12 months)
  Yes/No: study will be considered feasible if at least 80% of patients are satisfied.

SECONDARY OUTCOMES:
Compliance with completing the BEAUTIFY application | End of study (12 months)
  % of weeks where information is recorded out of the total number of weeks
Patient quality of life following surgery | Baseline
  European Organisation For Research And Treatment Of Cancer Quality of Life of Cancer Patients (EORTC QLQ C30): score of 1-7 for each item
Patient quality of life following surgery | 1 month
  EORTC QLQ C30: score of 1-7 for each item
Patient quality of life following surgery | 3 months
  EORTC QLQ C30: score of 1-7 for each item
Patient quality of life following surgery | 6 months
  EORTC QLQ C30: score of 1-7 for each item
Satisfaction of patients with their care | 1 month
  EORTC PATSAT-C33: score 0-100
Satisfaction of patients with their care | 3 months
  EORTC PATSAT-C33: score 0-100
Satisfaction of patients with their care | 6 months
  EORTC PATSAT-C33: score 0-100
Rate of post-operative complications | 6 months
  % patients with a complication noted in medical file
Type of post-operative complications | 6 months
  List of the complications affected patients as noted in medical file
Readmission rate for surgical or medical reason | 6 months
  % patients readmitted
Return to work and/or social activities | 1 year
  Date: Patients contacted by email or telephone

CONTACTS AND LOCATIONS:
Overall Officials: Frédéric Fiteni, Principal Investigator — CHU de Nimes
Locations (1):
- CHU de Nîmes, Nîmes, France